CLINICAL TRIAL: NCT00128401
Title: Effect of D-Cycloserine on Treatment of Social Phobia
Brief Title: Use of an Antibiotic as an Enhancer for the Treatment of Social Phobia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 050198; 05-M-0198
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-04

CONDITIONS: Phobic Disorders; Anxiety; Social Phobia
Keywords: Cognitive; Behavioral; Adolescent; Therapy; Extinction; Social Phobia
MeSH Terms: conditions — Phobic Disorders; Anxiety Disorders; Phobia, Social; Behavior | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- D-Cycloserine (Active Comparator): An antibiotic, d-cycloserine (DCS) was given to one group and the group is evaluated to see if the drug boosts the effectiveness of cognitive behavior therapy (CBT) for social anxiety.
  Interventions: Drug: D-Cycloserine
- Placebo (Placebo Comparator): Another group was given the placebo and tested for effectiveness of cognitive behavior therapy (CBT) for social anxiety.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-Cycloserine
  Arms: D-Cycloserine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study examines whether an antibiotic, d-cycloserine (DCS), boosts the effectiveness of cognitive behavior therapy (CBT) for social anxiety. CBT has been shown to be effective for the treatment of social anxiety in children and adults, but even after treatment, approximately 40% may remain diagnosable. The antibiotic DCS has been shown to enhance the type of learning that is promoted by exposure therapy, a main component of CBT. This study will test whether DCS can improve the effectiveness of CBT for social anxiety.

All participants will receive 12 weekly CBT sessions. In addition to receiving the CBT, participants will be randomly assigned (similar to a coin toss) to receive either DCS or a placebo (sugar pill). The pill will be taken 1-2 hours prior to each of the 12 CBT sessions. The pill is taken only on the 12 therapy days.

Prior to receiving treatment, participants will be asked to:

* participate in interviews to assess diagnosis and how they are doing including mood, degree of nervousness and behavior
* have a physical examination, a urine test, and an electrocardiogram (EKG)
* undergo tests involving problem-solving and memory
* prepare and present a speech to a "virtual audience" using virtual reality goggles
* undergo functional magnetic resonance imaging (fMRI) while performing tasks that involve looking at pictures, remembering things, testing reaction times, and making simple choices

Those who have not improved by the end of the study will be offered standard antianxiety medication treatment for 1 to 3 months. If a participant does not wish to take medication, study clinicians will help him/her locate psychological care in the community. Participants will be asked to complete a follow-up assessment 3 months after their last CBT session.

DETAILED DESCRIPTION:
Social phobia afflicts between 3%-15% of the US population. As such, it is a particularly common debilitating psychiatric disorder. Like many anxiety disorders, social phobia typically arises during adolescence. Treatment has consisted of medication or cognitive behavioral therapy (CBT). Selective Serotonin Reuptake Inhibitors (SSRIs) represent the first-line pharmacological treatment both in adults as well as adolescents (APA Treatment Guidelines 2004). Similarly, CBT significantly improves outcome in both age groups. This treatment consists of psychoeducation, exposure therapy, and cognitive restructuring. While both treatments produce clinically meaningful benefits, most patients exhibiting positive responses to these treatments continue to exhibit marked residual symptoms, if not full-blown anxiety disorders. Thus, there is great need for treatment advances.

Intense fear of social scrutiny represents a core component of social phobia, and extinction of this fear represents the goal of exposure therapy during CBT (Cohn and Hope). Finding treatments that facilitate extinction is of paramount importance. In animals, extinction involves an active learning process that is blocked by glutamatergic NMDA antagonists and facilitated by NMDA agonists. Specifically, administration of D-cycloserine (DCS), a partial agonist at the glycine modulatory site on the NMDA receptor, produces a dose-dependent facilitation of extinction in the rat. As such, DCS might facilitate extinction during exposure-based CBT. Indeed, Ressler (Ressler et al 2004) recently reported preliminary data from a clinical trial supporting this hypothesis.

We will examine the degree to which DCS treatment can augment the clinical response in social phobia to CBT-exposure-based therapy. Specifically, we will study two groups of individuals with social phobia, both of whom will receive CBT. One group will receive placebo; a second group will receive 50 mg of D-cycloserine 1-2 hours before each exposure therapy session. We hypothesize that compared to placebo, DCS will produce greater reductions in social anxiety symptoms following CBT treatment. Finally, given that chronic social anxiety disorder virtually always begins during childhood, it is particularly vital to develop early interventions for the disorder. Accordingly, our trial will examine both adolescents and adults with the disorder.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subjects between 8 yrs of age (preadolescents) and under 55 yrs of age.
  2. Subjects medically healthy.
  3. Able to give informed consent.
  4. Not on psychotropic meds for a minimum of 6 weeks for fluoxetine; a minimum of 1 week for PRN benzodiazepines and beta blockers, and a minimum of 3 weeks for all other psychotropic meds.
  5. Subjects diagnosed with DSM IV symptoms of social phobia, generalized or specific type.

EXCLUSION CRITERIA:

1. Current major depressive disorder.
2. Lifetime diagnosis of psychotic disorder, bipolar disorder, eating disorder, mental retardation, substance or alcohol dependence (other than nicotine); active suicidal ideation.
3. Current or lifetime history of a neurological disorder (other than tic disorders, febrile seizures of infancy), seizure disorder.
4. Any unstable medical condition.
5. Use of any psychoactive substance in the past 30 days.

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2005-08; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Cameron, C.R.N.P., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Alstrom JE, Nordlund CL, Persson G, Harding M, Ljungqvist C. Effects of four treatment methods on social phobic patients not suitable for insight-oriented psychotherapy. Acta Psychiatr Scand. 1984 Aug;70(2):97-110. doi: 10.1111/j.1600-0447.1984.tb01187.x. PMID 6148843
- [Background] Butler G, Cullington A, Munby M, Amies P, Gelder M. Exposure and anxiety management in the treatment of social phobia. J Consult Clin Psychol. 1984 Aug;52(4):642-50. doi: 10.1037//0022-006x.52.4.642. No abstract available. PMID 6147366
- [Background] D'Souza DC, Gil R, Cassello K, Morrissey K, Abi-Saab D, White J, Sturwold R, Bennett A, Karper LP, Zuzarte E, Charney DS, Krystal JH. IV glycine and oral D-cycloserine effects on plasma and CSF amino acids in healthy humans. Biol Psychiatry. 2000 Mar 1;47(5):450-62. doi: 10.1016/s0006-3223(99)00133-x. PMID 10704956
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-M-0198.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants were enrolled, but not assigned to treatment.
Groups:
- D-cycloserine: Subjects were randomized to receive cognitive behavioral therapy with augmentation of D-cycloserine 50 mg administered on day of therapy session. All subjects underwent the same intake procedures and the same procedures for the assessments for baseline severity. Morever all subjects began the same psychotherapy procedures using cognitive behavioral therapy. After cognitive behavioral therapy was initiated subjects were randomized into a 1:1 ratio by the NIH pharmacy to enter either continued therapy with placebo or continued therapy with the active agent.
- Placebo: Subjects were randomized to receive cognitive behavioral therapy with augmentation of placebo administered on day of therapy session.
  All subjects underwent the same intake procedures and the same procedures for the assessments for baseline severity. Morever all subjects began the same psychotherapy procedures using cognitive behavioral therapy. After cognitive behavioral therapy was initiated subjects were randomized into a 1:1 ratio by the NIH pharmacy to enter either continued therapy with placebo or continued therapy with the active agent.
Period: Overall Study
Arm/Group | D-cycloserine | Placebo
Started | 20 | 19
Completed | 14 | 15
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Population: The baseline mean and SD for CGI outcome measure was captured for 42 subjects only. The baseline mean and SD for LSAS outcome measure was captured for 40 subjects. Only 39 subjects were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 7 | 14
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 12 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 20 | 17 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 12 | 12 | 24
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Clinical Global Impressions (CGI) - baseline [Mean (Standard Deviation); unit: Units on a scale] — Symptom severity and improvement was assessed using the Clinical Global Impressions scale (CGI). It is a 2-item clinician-administered instrument that measures severity and improvement. One item characterizes subjects at baseline and at each post-baseline visit, based on severity. This is the CGI-S scale. This scale ranges from a score of 1 (normal, not all ill) to 7 (among the most extremely ill patients). The second item, the primary efficacy measure, is only rated after baseline, to quantify the amount of change. This ranges from 1 (completely recovered) to 8 (much worse).
  Units on a scale | 4.35 (0.587) | 4.278 (0.576) | 4.286 (0.554)
Liebowitz Social Anxiety Scale (LSAS) - baseline [Mean (Standard Deviation); unit: Units on a scale] — Social anxiety symptoms were assessed using the Liebowitz Social Anxiety Scale (LSAS). It is a 24-item self-report instrument that measures overall social anxiety fear and avoidance symptoms. This is the baseline assessment. The 24 items are each rated twice, from a "0" to "3" scale, with "0" indicated no level of symptom and "3" indicating a high level of the system. One rating is for anxiety, and the other is for avoidance. Thus, the lowest possible score is 0, and the highest possible score is 144. The total score represents the simple sum of all 48 ratings.
  Units on a scale | 89.9 (27.028) | 75.588 (25.063) | 83.725 (25.910)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Improvement (CGI-S) Scale
Description: Symptom severity and improvement was assessed using the Clinical Global Impressions scale (CGI). It is a 2-item clinician-administered instrument that measures the patients' illness severity and global improvement. The minimum value for the CGI is 1=Normal, not at all ill and the maximum value is 7=Among the most extremely ill patients.
Time Frame: 12 weeks post baseline
Population: The analyses included only those subjects who were assigned to the DCS condition and placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 4.167 (0.577) | 3.833 (0.835)

2. Secondary Outcome: Liebowitz Social Anxiety Scale (LSAS)
Description: Social anxiety symptoms were assessed using the Liebowitz Social Anxiety Scale (LSAS). It is a 24-item self-report instrument that measures overall social anxiety fear and avoidance symptoms. This is the baseline assessment. The 24 items are each rated twice, from a "0" to "3" scale, with "0" indicated no level of symptom and "3" indicating a high level of the system. One rating is for anxiety, and the other is for avoidance. Thus, the lowest possible score is 0, and the highest possible score is 144. The total score represents the simple sum of all 48 ratings.
Time Frame: 12 weeks post baseline
Population: The analyses included only those subjects who were assigned to the DCS condition and placebo
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 12 | 13
units on a scale | 74.417 (28.804) | 56.154 (20.066)

ADVERSE EVENTS:
Arm/Group | D-cycloserine | Placebo | Not Assigned
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/9
Other Adverse Events (participants affected / at risk) | 10/20 | 12/19 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | D-cycloserine (N=20) | Placebo (N=19) | Not Assigned (N=9)
Congenital, familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 0 | 1 | 0
Endocrine disorders - Other, specify (Thyroid problem) (Endocrine disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Fever (General disorders) | 0 | 1 | 0
Flu like symptoms (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specify (Cold symptoms) (General disorders) | 1 | 4 | 0
General disorders and administration site conditions - Other, specify (Cold) (General disorders) | 0 | 1 | 0
General disorders and administration site conditions - Other, specify (congestion) (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specify (missed medication) (General disorders) | 3 | 1 | 0
General disorders and administration site conditions - Other, specify (missed treatment session) (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specify (Runny nose) (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specify (stopped medication) (General disorders) | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (tail bone cyst) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (broken left arm) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 2 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0
Uterine pain (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Pruritus (Itching from broken arm) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The baseline mean and SD for CGI outcome measure was captured for 42 subjects only. The baseline mean and SD for LSAS outcome measure was captured for 40 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes